CLINICAL TRIAL: NCT01602185
Title: Antagonists NMDA in Relay to Ketamine in Neuropathic Pain
Brief Title: Study of NMDA Antagonists and Neuropathic Pain
Acronym: NMDA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Dr Malou Navez, Pain Clinic, Saint-Etienne Hopital (Unknown); Dr Marc Sorel, Pain Clinic, Nemours Hospital (Unknown); Dr Anne-Margot Duclot, Pain Clinic, Paris Rotschild Hospital (Unknown); Dr Monique Belon, Pain Clinic, Aurillac Hospital (Unknown); Dr Marie-Christine Crosmary/Dr Renato Colamarino, Pain Clinic, Vichy Hospital (Unknown); Dr Mohamed El Ayadi, Pain Clinic, Issoire Hospital (Unknown); Dr Géraldine Brumauld de Montgazon, Pain Clinic, La Rochelle Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0112
Record Dates: First submitted 2012-01-27; First posted 2012-05-18 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Neuropathic Pain
Keywords: NMDA (N-Methyl-D-Aspartate) antagonists; ketamine; memantine; dextromethorphan; Neuropathic pain
MeSH Terms: conditions — Neuralgia | interventions — Dextromethorphan; Memantine; Amyloid beta-Protein Precursor; Lactose

ARMS (3):
- memantine (Experimental): The aim of this study is to evaluate if memantine or dextromethorphan gave in relay to ketamine maintains or induces a decrease of pain intensity
  Interventions: Drug: Memantine (drug used in Alzheimer's disease)
- dextromethorphan (Experimental): The aim of this study is to evaluate if memantine or dextromethorphan gave in relay to ketamine maintains or induces a decrease of pain intensity
  Interventions: Drug: Dextromethorphan (drug used like antitussive)
- placebo (Placebo Comparator): The aim of this study is to evaluate if memantine or dextromethorphan gave in relay to ketamine maintains or induces a decrease of pain intensity
  Interventions: Drug: Placebo (lactose)

INTERVENTIONS:
Drug: Dextromethorphan (drug used like antitussive) — The aim of this study is to evaluate if memantine or dextromethorphan gave in relay to ketamine maintains or induces a decrease of pain intensity
  Arms: dextromethorphan
Drug: Memantine (drug used in Alzheimer's disease) — The aim of this study is to evaluate if memantine or dextromethorphan gave in relay to ketamine maintains or induces a decrease of pain intensity
  Arms: memantine
Drug: Placebo (lactose) — The aim of this study is to evaluate if memantine or dextromethorphan gave in relay to ketamine maintains or induces a decrease of pain intensity
  Arms: placebo

SUMMARY:
The aim of this study is to evaluate if memantine or dextromethorphan gave in relay to ketamine maintains or induces a decrease of pain intensity.

In clinical, after ketamine cure, clinicians have often difficulties to treat patients in order to maintain analgesia or suggest another treatment if analgesia induced by ketamine was not effective, which occurs in one quarter of patients. It will be very useful for monitoring of painful patients evaluate if memantine or dextromethorphan could be an effective therapeutic alternative in neuropathic pain treatment.

DETAILED DESCRIPTION:
The aim of this study is to evaluate if memantine or dextromethorphan gave in relay to ketamine maintains or induces a decrease of pain intensity.

In clinical, after ketamine cure, clinicians have often difficulties to treat patients in order to maintain analgesia or suggest another treatment if analgesia induced by ketamine was not effective, which occurs in one quarter of patients. It will be very useful for monitoring of painful patients evaluate if memantine or dextromethorphan could be an effective therapeutic alternative in neuropathic pain treatment.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* patient suffering chronic neuropathic pain
* All chronic pain is retained except central or diabetic pain
* Answering patient at ketamine in pain treatment by investigator, and having already received ketamine
* Patient who completed before ketamine the following evaluation :

DN4, QCD, QDSA, PGIC questionnaires, HAD scale, Leed's sleep evaluation and SF36.

* Patient who completed at the end of treatment the following evaluation : numerical scale and PGIC
* Sufficient cooperation and understanding to comply to the requirements of study
* Acceptance to give a written concert
* Affiliation at system of French social security
* Inscription or acceptation of inscription at national register of voluntaries participant at research

Exclusion Criteria:

* Against-indication at memantine or dextromethorphan administration : hypersensitivity at active substance or excipients, hypertension, antecedent cerebrovascular accident, severe cardiac insufficiency
* Patient with medical or surgical antecedents
* Patient with progressive disease at balance of inclusion
* Patient treated by an IMAO
* Woman in childbearing age not using effective contraceptive method, pregnant or lactating woman
* Patient who participated in another clinical trial, located in exclusion period or received benefits > 4500 euros during 12 months before the beginning of trial
* Patient with cooperation and understanding insufficiency to comply to the requirements of protocol
* Patient with social protection
* No affiliation at system of French social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2016-09-07 (Actual)

PRIMARY OUTCOMES:
Measure of pain by numerical scale | at Day 30

SECONDARY OUTCOMES:
Measure of pain by numerical scale | at day 60 and at day 90
Patient Global Impression if Change (PGIC) | at day 30, at day 60 and at day 90
Leed's slip questionnaire | at day 30, at day 60 and at day 90
Questionnaire of quality of life SF 36 | at day 30, at day 60 and at day 90
DN4 scale | at day 30, at day 60 and at day 90
Neuropathic Pain Symptoms Inventory (NPSI) | at day 30, at day 60 and at day 90
Saint-Antoine questionnaire (QDSA) | at day 30, at day 60 and at day 90
HAD scale | at day 30, at day 60 and at day 90
Questionnaire of identification of pain (QCD) | at day 30, at day 60 and at day 90
Evaluation of cognitive impact (Cantab, Cambridge) | at day 30, at day 60 and at day 90

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle PICKERING, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Pickering G, Pereira B, Morel V, Tiberghien F, Martin E, Marcaillou F, Picard P, Delage N, de Montgazon G, Sorel M, Roux D, Dubray C. Rationale and design of a multicenter randomized clinical trial with memantine and dextromethorphan in ketamine-responder patients. Contemp Clin Trials. 2014 Jul;38(2):314-20. doi: 10.1016/j.cct.2014.06.004. Epub 2014 Jun 16. PMID 24948402